CLINICAL TRIAL: NCT05403827
Title: A Phase 3, Prospective, Double-masked, Randomized, Multi-center, Vehicle-controlled, Parallel-group, 12-week Administration and 40-week Extension Study Confirming the Efficacy and Safety of K-161 Ophthalmic Solution for the Treatment of Moderate to Severe Dry Eye Disease
Brief Title: A Study to Confirm the Efficacy and Safety of K-161 Ophthalmic Solution for Treatment of Moderate to Severe Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-161-3.01
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- K-161 (Experimental): K-161 Ophthalmic Solution
  Interventions: Drug: K-161
- Placebo (Placebo Comparator): Vehicle Solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-161 — K-161 Ophthalmic Solution
  Arms: K-161
Drug: Placebo — Vehicle Solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of K-161 ophthalmic solution for the treatment of moderate to severe dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at the time of Informed Consent
* Have a reported history of dry eye disease in both eyes and a history of eye drop use for dry eye symptom
* Meet all other inclusion criteria outlined in the clinical study protocol

Exclusion Criteria:

* Have any clinically significant ocular condition
* Have a history of corneal refractive surgery and/or any other ocular surgical procedure within 12 months
* Meet any other exclusion criteria outlined in the clinical study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey E. Belous, MD, PhD, Study Chair — Kowa Pharma Development Co.
Locations (51):
- United States (51):
  - The University of Alabama at Birmingham School of Optometry, Clinical Eye Research Center, Birmingham, Alabama
  - Trinity Research Group, Dothan, Alabama
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Citrus Valley Eyecare / Premiere Practice Management, LLC, Covina, California
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - Global Research Management, Glendale, California
  - Inland Eye Specialists, Hemet, California
  - United Medical Research Institute, Inglewood, California
  - Premiere Practice Management, LLC, Los Angeles, California
  - North Valley Eye Medical Group, Inc, Mission Hills, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Inc., Newport Beach, California
  - Pendleton Eye Center, Oceanside, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Sierra Clinical Trial Research Organization, Santa Ana, California
  - Premiere Practice Management, LLC, Torrance, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - Vision Institute, Colorado Springs, Colorado
  - Corneal Consultants of Colorado dba Colorado Eye Consultants, Littleton, Colorado
  - Segal Drug Trials, Delray Beach, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - International Research Center, Tampa, Florida
  - Dixophthal, PC., Albany, Georgia
  - Edwin Yoshio Endo, OD & Associates & Interns, ‘Aiea, Hawaii
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Jones Eye Clinic and Surgery Center, Sioux City, Iowa
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Midwest Vision Research Foundation at Pepose Vision Institute, Chesterfield, Missouri
  - Tauber Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Wellish Vision Institute, Las Vegas, Nevada
  - Asheville Eye Associates, Asheville, North Carolina
  - Oculus Research, Garner, North Carolina
  - Wake Forest Health Network, LLC, High Point, North Carolina
  - Insight Research Clinic, LLC dba EyeCare Professionals, Powell, Ohio
  - Conestoga Eye PC, Lancaster, Pennsylvania
  - Associates in Ophthalmology Ltd, West Mifflin, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, Smyrna, Tennessee
  - Keystone Research, Austin, Texas
  - Hill Country Eye Center, Cedar Park, Texas
  - Southwest Eye Institute, El Paso, Texas
  - Lake Travis Eye and Laser Center/Revolution Research, Lakeway, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - DCT-Shah Research, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Northern Virginia Ophthalmology Associates, Falls Church, Virginia
  - Virginia Eye Consultants, Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1 (Screening), eligible participants were provided single-masked run-in product (Vehicle) for self-administration in the morning and evening, for approximately 14 days. At Visit 2 (Baseline), participants who remained eligible for the study were randomized in a 1:1 ratio to double-masked IP (K-161 or Vehicle). Each participant provided voluntary informed consent before any study-specific assessments or procedures were performed.
Groups:
- K-161: K-161 topical Ophthalmic solution for 12 weeks
- Vehicle: Vehicle K-161 identical topical ophthalmic solution without active drug for 12 weeks
Period: 12 Week Primary
Arm/Group | K-161 | Vehicle
Started | 322 | 322
Completed | 253 (A single subject was randomized to the K-161 group but never received K-161 Ophthalmic Solution double-masked IP due to an adverse event) | 269
Not Completed | 69 | 53
Period: 52 Week Overall
Arm/Group | K-161 | Vehicle
Started | 122 (Proportion of participants from 12-Week primary period K-161 group continuing into 52-Week Overall period.) | 121 (Proportion of participants from 12-Week primary period vehicle group continuing into 52-Week Overall period.)
Completed | 67 | 75
Not Completed | 55 | 46

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the Safety Population in the 12-week Primary Period (SP12).
Groups:
- Total: Total of all reporting groups
Arm/Group | K-161 | Vehicle | Total
Number analyzed (Participants) | 321 | 322 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.88) | 60.0 (15.18) | 60.0 (14.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 234 | 467
  Male | 88 | 88 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 234 | 230 | 464
  Black or African American | 42 | 41 | 83
  Asian | 39 | 45 | 84
  Native Hawaiian | 0 | 1 | 1
  Other | 2 | 1 | 3
  Multiple | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in EDS (VAS) From Baseline to Day 85
Description: * Eye Dryness Score (EDS) on Visual analog scale (VAS)
  * Participant self rated level of severity where, 0 mm corresponds to "None" and 100 mm corresponds to "Worst Possible".
Time Frame: Baseline to Day 85
Population: The number of participants analyzed for the outcome measure may differ from the overall number of participants in each group. This discrepancy can be attributed to several factors, including:
  • Missing data: Some participants may have incomplete data due to factors such as missed visits, early withdrawal, or loss to follow-up.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 292 | 306
mm | -18.0 (25.10) | -19.4 (25.34)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.5019, Control-Based Mean Imputation

2. Primary Outcome: Change in Conjunctival Sum Fluorescein Staining Score From Baseline to Day 85 (Study Eye)
Description: * Assessed by expanded National Eye Institute (NEI) scale
  * Conjunctival sum will be assessed as the sum of points in 6 conjunctival zones, and each zone will be graded on a 5-point scale from 0 - no conjunctival staining to 4 - severe staining of the area (0.5 increments would be allowed)
  * Minimum is 0 and maximum is 24 for Conjunctival Sum Fluorescein Staining Score.
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 291 | 306
Score on a scale | -2.81 (3.661) | -3.25 (3.480)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.2028, Control-Based Mean Imputation

3. Secondary Outcome: Change From Baseline to Day 85 in Total Eye Sum Fluorescein Staining Score (Study Eye)
Description: * Assessed by expanded National Eye Institute (NEI) scale.
  * Total eye sum will be assessed as the sum of Corneal sum fluorescein staining score and conjunctival sum fluorescein staining score.
  * Minimum is 0 and maximum is 44 for Total Eye Sum Fluorescein Staining Score.
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 291 | 306
Score on a scale | -4.73 (5.693) | -5.44 (5.546)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.1914, Control-Based Mean Imputation

4. Secondary Outcome: Change From Baseline to Day 85 in Corneal Sum Fluorescein Staining Score (Study Eye)
Description: * Assessed by expanded National Eye Institute (NEI) scale.
  * Corneal sum will be assessed as the sum of points in 5 corneal zones, and each zone will be graded on a 5-point scale from 0 - no punctate stain in the area to 4 - Severe diffuse (coalescent) macropunctate stain of the area (0.5 increments would be allowed)
  * Minimum is 0 and maximum is 20 for Corneal Sum Fluorescein Staining Score
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 291 | 306
Score on a scale | -1.92 (2.905) | -2.19 (2.841)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.2512, Control-Based Mean Imputation

5. Secondary Outcome: Change From Baseline to Day 85 in Ocular Surface Disease Index Score (OSDI©)
Description: OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability.
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 292 | 306
Score on a scale | -14.12 (17.099) | -14.17 (17.594)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.7906, Control-Based Mean Imputation

6. Secondary Outcome: Change From Baseline to Day 85 in Schirmer's Test (Unanesthetized) (Study Eye)
Description: Length (mm) of the moistened area assessed by inserting a Schirmer test strip into the eye for 5 minutes to measure the production of tears.
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 291 | 306
mm | 2.4 (5.47) | 2.6 (5.25)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.5343, Control-Based Mean Imputation

7. Secondary Outcome: Change From Baseline to Day 85 in Tear Film Break-up Time (TFBUT) (Study Eye)
Description: The time (in seconds) taken for the first dry spot to appear on the cornea after a complete blink (with the aid of a slit-lamp).
Time Frame: Baseline to Day 85
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | K-161 | Vehicle
Number analyzed (Participants) | 291 | 305
Seconds | 0.580 (1.2089) | 0.520 (1.1989)
Statistical Analysis 1: Comparison: K-161 vs Vehicle; Test type: Superiority; p = 0.3757, Control-Based Mean Imputation

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Treatment emergent adverse events (TEAEs) were defined as AEs that began after the start of the double-masked IP dosing, or events that began before the start of the double-masked IP dosing and worsened in intensity after IP dosing began.
Groups:
- K-161 12-Week: The safety population included all participants treated in the 12-Week primary period (SP12) who received K-161 ophthalmic solution.
- Vehicle 12-Week: The safety population included all participants treated in the 12-Week primary period (SP12) who received vehicle solution.
- K-161 40-Week Extension: The analysis group consist of only subjects from the 40-Week extension period assigned to receive K-161 ophthalmic solution.
- Vehicle 40-Week Extension: The analysis group consist of only subjects from the 40-Week extension period assigned to receive Vehicle ophthalmic solution.
Arm/Group | K-161 12-Week | Vehicle 12-Week | K-161 40-Week Extension | Vehicle 40-Week Extension
All-Cause Mortality (participants affected / at risk) | 0/321 | 0/322 | 0/122 | 0/121
Serious Adverse Events (participants affected / at risk) | 3/321 | 2/322 | 1/122 | 2/121
Other Adverse Events (participants affected / at risk) | 32/321 | 0/322 | 0/122 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | K-161 12-Week (N=321) | Vehicle 12-Week (N=322) | K-161 40-Week Extension (N=122) | Vehicle 40-Week Extension (N=121)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-161 12-Week (N=321) | Vehicle 12-Week (N=322) | K-161 40-Week Extension (N=122) | Vehicle 40-Week Extension (N=121)
Instillation site pain (General disorders) | 32 | 0 | 0 | 0 — General Disorders and Administration Site Conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INSTITUTION/INVESTIGATOR may publish/present results after SPONSOR publication. Prior SPONSOR review protects confidential info & patentable material. Confidential info will be removed. Patentable findings may delay publication for patent filing. Acknowledgement of SPONSOR's support is at SPONSOR's option, with prior consent required for any SPONSOR reference.

DOCUMENTS (5):
  • Study Protocol: Initial (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT05403827/Prot_000.pdf
  • Study Protocol: Amendment 1 (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT05403827/Prot_001.pdf
  • Study Protocol: Amendment 2 (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05403827/Prot_002.pdf
  • Statistical Analysis Plan: Ver 1.0 (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT05403827/SAP_003.pdf
  • Statistical Analysis Plan: ver 1.0 Addendum (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT05403827/SAP_004.pdf